CLINICAL TRIAL: NCT01692535
Title: Multicenter Study Evaluating Video Laryngoscopes: The Swiss Video-Intubation Trial (SWIVIT I)
Brief Title: Evaluation of Video Laryngoscopes in Difficult Airway
Acronym: SWIVIT I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Lorenz Theiler, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 106/12
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Intubation; Difficult
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- GlideScope (Experimental): intubation
  Interventions: Procedure: Intubation
- Airtraq (Experimental): intubation
  Interventions: Procedure: Intubation
- McGrath MAC (Experimental): intubation
  Interventions: Procedure: Intubation
- King Vision (Experimental): intubation
  Interventions: Procedure: Intubation
- A.P. Advance (Experimental): intubation
  Interventions: Procedure: Intubation
- C-MAC (Experimental): intubation
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — Intubation with one of the six videolaryngoscopes

SUMMARY:
In this multicenter study the investigators are going to evaluate the use of six different videolaryngoscopes in patients undergoing elective surgery requiring general anesthesia with intubation. The investigators are hypothesizing that these six videolaryngoscopes will succeed for intubation at first attempt in at least 90% of all cases using a difficult airway simulation with extrication collars. As gold standard, a standard Macintosh blade is being used.

The study consists of 6 arms. Each arm includes 120 patients, sums up to a total of 720 patients.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery with general anesthesia requiring intubation
* >18years old
* ASA I-III

Exclusion Criteria:

* known or presumed difficult airway
* risk of pulmonary aspiration
* refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
First attempt intubation success rate | within 180 seconds

SECONDARY OUTCOMES:
side effects | 1h and 1 day after surgery
  sore throat, bleeding, dental injuries

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME FERC, Study Chair — University Dept Anesthesiology and Pain Therapy, University of Berne, Switzerland
Locations (3):
- Switzerland (3):
  - Bern University Hospital and University of Bern, Bern, Canton of Bern
  - Hopitaux Universitaires de Geneve HUG, Geneva, Canton of Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne, Canton of Vaud

REFERENCES:
- [Derived] Kleine-Brueggeney M, Greif R, Schoettker P, Savoldelli GL, Nabecker S, Theiler LG. Evaluation of six videolaryngoscopes in 720 patients with a simulated difficult airway: a multicentre randomized controlled trial. Br J Anaesth. 2016 May;116(5):670-9. doi: 10.1093/bja/aew058. PMID 27106971
- [Derived] Theiler L, Hermann K, Schoettker P, Savoldelli G, Urwyler N, Kleine-Brueggeney M, Arheart KL, Greif R. SWIVIT--Swiss video-intubation trial evaluating video-laryngoscopes in a simulated difficult airway scenario: study protocol for a multicenter prospective randomized controlled trial in Switzerland. Trials. 2013 Apr 4;14:94. doi: 10.1186/1745-6215-14-94. PMID 23556410